CLINICAL TRIAL: NCT06605378
Title: A Cross-Sectional, Observational Study of the Prevalence of Adenoviral-Specific Antibodies and Inflammatory Cytokines in Participants With Chronic Granulomatous Disease
Brief Title: Prevalence of Antibodies and Cytokines in Participants With Chronic Granulomatous Disease
Status: Recruiting | Type: Observational
Sponsor: Ensoma (Industry)
Responsible Party: Sponsor
Other Study IDs: EN-374-100
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Granulomatous Disease (CGD)
Keywords: CGD; X-CGD; Chronic Granulomatous Disease; Granulomatous Disease, Chronic; Autosomal Recessive Chronic Granulomatous Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is designed to assess the prevalence of specific antibodies and inflammatory cytokines in adult and pediatric participants with CGD.

DETAILED DESCRIPTION:
In this observational study, blood samples will be collected from adult and pediatric patients with CGD. The level of circulating adenovirus antibodies and inflammatory cytokines will be measured to characterize the prevalence of these markers in this population.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have been diagnosed with CGD based on the referring physician's confirmation that NADPH oxidase activity is ≤5% (i.e., the percentage of dihydrorhodamine-positive [DHR+] cells is ≤5% by flow cytometry) OR based on confirmed pathogenic mutation in a CGD associated gene (CYBB, CYBA, NCF1, NCF2, NCF4, or CYBC1).
* The participant or the participant's legally authorized guardian or representative (if applicable) must be capable of giving signed informed consent.
* The participant (with assistance from the participant's legally authorized guardian/representative or primary caregiver, if applicable) must be capable of complying with the requirements and restrictions listed in the protocol and informed consent form (ICF).

Exclusion Criteria:

* The participant has undergone an allogeneic bone marrow transplant or investigational gene therapy.
* The participant is unable to comply with the sample collection procedure based on investigator judgment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with CGD
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total adenoviral-specific antibody (TAb) titer | 1 Day
  Level of total adenoviral-specific antibody in blood
Adenoviral-specific neutralizing antibody (NAb) titer | 1 Day
  Level of adenoviral-specific neutralizing antibodies in blood

SECONDARY OUTCOMES:
Circulating inflammatory cytokine levels | 1 Day
  Level of inflammatory cytokines in blood

CONTACTS AND LOCATIONS:
Locations (52):
- United States (50):
  - Home-based telemedicine, Montgomery, Alabama
  - Home-based telemedicine, Phoenix, Arizona
  - Home-based telemedicine, Little Rock, Arkansas
  - Home-based telemedicine, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Home-based telemedicine, Denver, Colorado
  - Home-based telemedicine, Hartford, Connecticut
  - Home-based telemedicine, Dover, Delaware
  - Home-based telemedicine, Washington D.C., District of Columbia
  - Home-based telemedicine, Tallahassee, Florida
  - Home-based telemedicine, Atlanta, Georgia
  - Home-based telemedicine, Boise, Idaho
  - Home-based telemedicine, Springfield, Illinois
  - Home-based telemedicine, Indianapolis, Indiana
  - Home-based telemedicine, Des Moines, Iowa
  - Home-based telemedicine, Topeka, Kansas
  - Home-based telemedicine, Frankfort, Kentucky
  - Home-based telemedicine, Baton Rouge, Louisiana
  - Home-based telemedicine, Augusta, Maine
  - Home-based telemedicine, Annapolis, Maryland
  - Home-based telemedicine, Boston, Massachusetts
  - Home-based telemedicine, Lansing, Michigan
  - Home-based telemedicine, Saint Paul, Minnesota
  - Home-based telemedicine, Jackson, Mississippi
  - Home-based telemedicine, Jefferson City, Missouri
  - Home-based telemedicine, Helena, Montana
  - Home-based telemedicine, Lincoln, Nebraska
  - Home-based telemedicine, Carson City, Nevada
  - Home-based telemedicine, Concord, New Hampshire
  - Home-based telemedicine, Trenton, New Jersey
  - Home-based telemedicine, Santa Fe, New Mexico
  - Home-based telemedicine, Albany, New York
  - Science 37, Inc, Morrisville, North Carolina
  - Home-based telemedicine, Bismarck, North Dakota
  - Home-based telemedicine, Columbus, Ohio
  - Home-based telemedicine, Oklahoma City, Oklahoma
  - Home-based telemedicine, Salem, Oregon
  - Home-based telemedicine, Harrisburg, Pennsylvania
  - Home-based telemedicine, Providence, Rhode Island
  - Home-based telemedicine, Columbia, South Carolina
  - Home-based telemedicine, Pierre, South Dakota
  - Home-based telemedicine, Nashville, Tennessee
  - Home-based telemedicine, Austin, Texas
  - Home-based telemedicine, Salt Lake City, Utah
  - Home-based telemedicine, Montpelier, Vermont
  - Home-based telemedicine, Richmond, Virginia
  - Home-based telemedicine, Olympia, Washington
  - Home-based telemedicine, Charleston, West Virginia
  - Home-based telemedicine, Madison, Wisconsin
  - Home-based telemedicine, Cheyenne, Wyoming
- United Kingdom (2):
  - Great Ormond Street Hospital for Children, London
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No